CLINICAL TRIAL: NCT02004925
Title: Accuracy of Ultrasonography for the Diagnosis of Pneumoperitoneum in the Emergency Department
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Peiman Nazerian, Medical Doctor Emergency Medicine, Azienda Ospedaliero-Universitaria Careggi
Other Study IDs: 070675
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Pneumoperitoneum
Keywords: pneumoperitoneum; free peritoneal air; ultrasonography
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pneumoperitoneum: Patients with a diagnosis of pneumoperitoneum by CT or surgery
- no pneumoperitoneum: patients with acute abdominal pain with a diagnosis other than pneumoperitoneum in whom pneumoperitoneum was excluded by CT or surgery

SUMMARY:
Pneumoperitoneum could be due to life threatening conditions and its quickly diagnosis is important in the emergency department (ED). Signs and symptoms are non-specific and radiography has low accuracy in the acute setting. Computed tomography (CT) is considered the gold standard, however it is not a cost-effective option in the vast population of patients with abdominal pain. Ultrasonography is able to detect as little as 2 ml of free air, however diagnostic accuracy of ultrasonography remains unclear. This study evaluates the accuracy of ultrasonography for the diagnosis of pneumoperitoneum, the most accurate abdominal scan and the most accurate echographic sign for the detection of free air.

Methods Consecutive patients presenting to ED for acute abdominal pain and with a diagnosis of pneumoperitoneum at CT or at surgery (study group) and a similar number of patients without a diagnosis of pneumoperitoneum (control group) undergo abdominal ultrasonography in a standardized protocol that include 10 scans for each patient registered on a video of 5 seconds. The videos are randomly reviewed by 4 sonographers and by 2 physicians with no experience in ultrasonography blind to final diagnosis and to all clinical data with the aim of detecting for each scan pneumoperitoneum. Accuracy of ultrasonography for the diagnosis of pneumoperitoneum will be calculated considering CT or surgery as gold standard. Furthermore intra and interobserver agreement and the accuracy of each ultrasonographic sign and scan will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* All patients more than 18 years with acute abdominal pain

Exclusion Criteria:

* Refused consent
* Less than 18 years old
* Not possible to perform ultrasonography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients more than 18 years presenting to emergency departments with acute abdominal pain and clinical suspected pneumoperitoneum
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Accuracy of ultrasonography for the diagnosis of pneumoperitoneum | No follow-up for the included patients. Outcome is measured one month after the end of recruitment
  CT or surgery are considered the gold standard for the diagnosis of pneumoperitoneum

SECONDARY OUTCOMES:
Accuracy of each scan and of each sonographic sign for the diagnosis of pneumoperitoneum | No follow-up for the included patients. Outcome is measured one month after the end of recruitment

OTHER OUTCOMES:
Inter and intraobserver agreement between reviewers | No follow-up for the included patients. Outcome is measured one month after the end of recruitment
  Concordance between the reviewers of the ultrasonographic videos for pneumoperitoneum diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Grifoni, MD, Study Chair — Director of Emergency Department AUO Careggi
Locations (1):
- Emergency Department Azienda Ospedaliera Universitaria Careggi, Florence, Italy

REFERENCES:
- [Derived] Nazerian P, Tozzetti C, Vanni S, Bartolucci M, Gualtieri S, Trausi F, Vittorini M, Catini E, Cibinel GA, Grifoni S. Accuracy of abdominal ultrasound for the diagnosis of pneumoperitoneum in patients with acute abdominal pain: a pilot study. Crit Ultrasound J. 2015 Dec;7(1):15. doi: 10.1186/s13089-015-0032-6. Epub 2015 Oct 6. PMID 26443344